CLINICAL TRIAL: NCT04114994
Title: Longitudinal Cognitive Assessment by BoCA
Acronym: BoCA
Status: Recruiting | Type: Observational
Sponsor: Alzheimer's Light LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BoCA001
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Vascular Dementia; Frontotemporal Dementia; Parkinson Disease; Multiple Sclerosis; TBI
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia, Vascular; Frontotemporal Dementia; Parkinson Disease; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Alzheimer's Disease
  Interventions: Diagnostic Test: Boston Cognitive Assessment (BoCA)
- Mild Cognitive Impairment
  Interventions: Diagnostic Test: Boston Cognitive Assessment (BoCA)
- Frontotemporal Dementia
  Interventions: Diagnostic Test: Boston Cognitive Assessment (BoCA)
- Vascular Dementia
  Interventions: Diagnostic Test: Boston Cognitive Assessment (BoCA)
- Parkinson Disease
  Interventions: Diagnostic Test: Boston Cognitive Assessment (BoCA)
- Traumatic Brain Injury (TBI)
  Interventions: Diagnostic Test: Boston Cognitive Assessment (BoCA)
- Multiple Sclerosis
  Interventions: Diagnostic Test: Boston Cognitive Assessment (BoCA)
- No diagnosis
  Interventions: Diagnostic Test: Boston Cognitive Assessment (BoCA)

INTERVENTIONS:
Diagnostic Test: Boston Cognitive Assessment (BoCA) — The Boston Cognitive Assessment (BoCA) is a self-administered online test intended for longitudinal cognitive monitoring. BoCA uses random not-repeating tasks to minimize learning effects. BoCA was developed to evaluate the effects of treatment in longitudinal clinical trials and available gratis to individuals and professionals.
  BoCA includes eight subtests in the following domains: Memory/Immediate Recall, Memory/Delayed Recall, Executive function/ Visuospatial, Executive function/ Mental rotation, Attention, Mental math, Language/Prefrontal Synthesis, and Orientation. The maximum total score is 30. Higher score indicates better cognitive performance.
  After BoCA is completed, the domain scores and total score are provided immediately. Users will also receive an email with the link to the full report with progress charts.

SUMMARY:
The Boston Cognitive Assessment (BoCA) is a self-administered online test intended for longitudinal cognitive monitoring. BoCA uses random not-repeating tasks to minimize learning effects. BoCA was developed to evaluate the effects of treatment in longitudinal clinical trials and available gratis to individuals and professionals.

DETAILED DESCRIPTION:
The Boston Cognitive Assessment (BoCA) is a self-administered online test intended for longitudinal cognitive monitoring. BoCA uses random not- repeating tasks to minimize learning effects. BoCA was developed to evaluate the effects of treatment in longitudinal clinical trials and available gratis to individuals and professionals.

BoCA includes eight subtests in the following domains: Memory/Immediate Recall, Memory/Delayed Recall, Executive function/ Visuospatial, Executive function/ Mental rotation, Attention, Mental math, Language/Prefrontal Synthesis, and Orientation. The maximum total score is 30. Higher score indicates better cognitive performance.

After BoCA is completed, the domain scores and total score are provided immediately. Users will also receive an email with the link to the full report with progress charts.

The BoCA evaluation can help doctors figure out if an underlying condition is causing a patient's cognitive decline. Many treatable conditions such as sleep disorders, mood problems, heavy metal accumulation, as well as lack of movement and social interactions can affect memory and thinking.

Our goal is to reduce barriers for patients to receive the testing that may benefit their treatment and health through the use of digital technology.

ELIGIBILITY:
Inclusion Criteria:

age 50 or older

Exclusion Criteria:

younger than 50 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to the American Academy of Neurology, nearly 7% of people in their early 60s worldwide have mild cognitive impairment, while the condition affects 38% of people ages 85 and older.
  The BoCA evaluation can help doctors figure out if an underlying condition is causing a patient's cognitive decline. Many treatable conditions such as sleep disorders, mood problems, heavy metal accumulation, as well as lack of movement and social interactions can affect memory and thinking.
  Our goal is to reduce barriers for patients to receive the testing that may benefit their treatment and health through the use of digital technology.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Boston Cognitive Assessment (BoCA) | through study completion, an average of 1 year
  The Boston Cognitive Assessment (BoCA) is a self-administered online test intended for longitudinal cognitive monitoring. BoCA uses random not-repeating tasks to minimize learning effects. BoCA was developed to evaluate the effects of treatment in longitudinal clinical trials and available gratis to individuals and professionals.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrey Vyshedskiy, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Foster NL, Bondi MW, Das R, Foss M, Hershey LA, Koh S, Logan R, Poole C, Shega JW, Sood A, Thothala N, Wicklund M, Yu M, Bennett A, Wang D. Quality improvement in neurology: Mild cognitive impairment quality measurement set. Neurology. 2019 Oct 15;93(16):705-713. doi: 10.1212/WNL.0000000000008259. Epub 2019 Sep 18. No abstract available. PMID 31534026
- See also: BoCA website — http://boca.alz.life